CLINICAL TRIAL: NCT06267508
Title: Increasing Neonatal HIV Test and Treat to Maximize the Long-Term Impact on Infant Health and Novel Infant Antiretroviral Treatment
Acronym: LIFE2Scale
Status: Recruiting | Type: Observational
Sponsor: Michael Hoelscher (Other)
Collaborators: National Institute for Medical Research (NIMR) - Mbeya Medical Research Centre (MMRC) (Unknown); Instituto Nacional de Saúde (INS), Ministério da Saúde (Unknown); University of Liverpool (Other)
Responsible Party: Sponsor-Investigator, Michael Hoelscher, Director, Division of Infectious Diseases and Tropical Medicine, University Hospital, LMU Munich,, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Other Study IDs: LMU-IMPH-LIFE2Scale
Record Dates: First submitted 2024-01-24; First posted 2024-02-20 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Vertical Human Immunodeficiency Virus Transmission; HIV Infection Pediatric; Infant Death; Infant Morbidity; Infant, Newborn, Diseases
Keywords: Prevention of Vertical HIV Transmission (PVHT); Infant HIV Prophylaxis; Early Infant HIV Diagnosis; Infant Antiretroviral Treatment
MeSH Terms: conditions — Infant Death; Infant, Newborn, Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort A: HIV-exposed infants and their mothers enrolled in the study
  Interventions: Procedure: Maternal HIV viral load testing at delivery for VHT risk assessment
- Cohort B: HIV-positive infants, identified in the first 12 weeks, and their mothers will be rolled over from Cohort A to Cohort B for long-term follow-up for up to 12 months.

INTERVENTIONS:
Procedure: Maternal HIV viral load testing at delivery for VHT risk assessment — Maternal HIV viral load testing will be performed for all mothers enrolled in the study at delivery. Results will be used along with WHO-defined clinical criteria to determine risk status for VHT. The intervention also includes personnel to support the additional testing volume and management of high-risk cases and eHealth solutions for communication of test results between health facilities.
  Groups: Cohort A

SUMMARY:
This study aims to improve HIV healthcare services for mothers living with HIV and their newborns in Tanzania and Mozambique. The main questions it aims to answer are: 1) does enhancing screening with maternal HIV viral load monitoring at delivery identify more mother-child pairs at high-risk for HIV vertical transmission? and 2) are high-risk infants linked to appropriate prevention and care? The study will expand access to HIV testing services to more rural settings using a hub-and-spoke referral system.

DETAILED DESCRIPTION:
The UN Sustainable Development Goals set the ambitious goal to eliminate new paediatric HIV infections by 2030. Between 2010 and 2020, new HIV infections among children declined by more than 50%. This decline demonstrates the goal is achievable, but the loss of momentum in recent years indicates a need for further improvements. Results from the previous LIFE study conducted in Mozambique and Tanzania demonstrated that identifying HIV-infection in neonates and starting HIV treatment as early as birth is feasible and may reduce infant death and severe disease. However, this study also demonstrated that it is difficult to administer infant HIV treatments due to poor palatability of the infant drug formulation, socio-behavioural constraints for mothers, and care linkage challenges. This resulted in poor treatment adherence and efficacy (as measured by HIV suppression rates in the blood).

The investigators propose to expand and optimize treatment and prevention interventions for mothers living with HIV and their newborns and translate previous research findings into policy and practice, with a focus on primary healthcare to reduce access inequities in rural areas. The study aims to scale-up of tools used for vertical HIV transmission risk screening affiliated with immediate, risk-based HIV test & treat procedures. Testing for high-risk case detection will be implemented in a hub-and-spoke model, where smaller, less well-equipped health facilities refer samples to nearby larger health facilities for diagnostic testing, ensuring rural communities have access to the interventions. The investigators will also provide personnel support for scale-up of high-risk case detection and high-risk infant care management. Furthermore, all high-risk mother-baby pairs will receive enhanced counselling services. eHealth tools for electronic result sharing across health facilities will be part of our package of interventions.

The investigators will evaluate the impact of the intervention package described above on key prevention of vertical HIV transmission (PVHT) program indicators (e.g., percentage of high-risk newborns immediately tested for HIV, percentage of newborns with HIV immediately started on treatment) in a stepped-wedge, cluster-randomized study. The investigators will also conduct a cost-effectiveness analysis of the intervention package. Furthermore, the investigators will conduct interviews and use self-reported questionnaires by the participants and site staff to better understand the socio-economic and behavioural factors contributing to high-risk classification.

For HIV-positive babies, the investigators will assess the impact of a novel HIV drug used for newborns, i.e. Dolutegravir (DTG), on health outcomes. The investigators will also characterize the impact of transmitted and acquired genotypic drug resistance, as well as transmitted viral strains, towards neutralization against established and novel broadly neutralizing antibodies. This information will be used to inform future prevention and treatment strategies for HIV-exposed newborns.

All mothers of HIV-positive babies taking part in this study will continue to have access to enhanced counselling and care support throughout the study, and the investigators will collect information on socio-behavioural factors influencing treatment outcomes to understand challenges related to infant HIV treatment.

This study will be performed by an established consortium of interdisciplinary African and European experts, closely collaborating with health authorities and policy makers, thus ensuring effective and sustainable implementation, programmatic stewardship, and global access to the proposed complex intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary and informed consent of the mother for her own study participation (if applicable);
2. Voluntary and informed consent of the legal guardian of the child for participation of the child in the study;
3. Mothers/legal guardians ≥18 years of age;
4. Documented maternal HIV infection;
5. Willingness to consent to HIV testing for the child and herself (or just her child); and
6. Willingness to consent to active tracing including home tracing.

   Exclusion Criteria:
7. Deficiency in the mother, rendering it difficult, if not impossible, for her or her infant to take part in the study or understand the information provided to her.
8. Having delivered more than 72h (3 days) ago;
9. Prisoners;
10. Women presenting with an emergency requiring immediate medical assistance if not resolved at study inclusion;
11. Stillbirths;
12. Infant requiring emergency care (e.g. immediate or rapid occurring life threatening conditions, resuscitation, prolonged obstetric related intensive care, severe jaundice) or born with severe malformation;
13. If within the discretion of the investigator based on recommendation of the gynaecologist or paediatrician in charge study participation would possibly add not acceptable risk or burden to the mother or infant (e.g. significant congenital malformation, health deficiencies, very low birth weight less than 1500g); or
14. Unlikely to comply with protocol as judged by the principal investigator or his designate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Mothers living with HIV presenting for delivery at included health facilities
Study Population: Pregnant women living with HIV and their exposed infants recruited at maternity clinics in Mozambique and Tanzania. The investigators expect to recruit 4000-6000 mother-child pairs in 12 months, or 56-71 mother-child pairs per cluster-randomization period (7 weeks) into Cohort A.
  Assuming 12-week VHT rates of 2.5% and 1% VHT rates in Mozambique and Tanzania respectively, the investigators expect to roll-over approximately 105 HIV positive infants (75 in Mozambique and 30 in Tanzania) from both countries into Cohort B.
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of HIV-exposed infants correctly identified as low- or high-risk and receiving birth EID testing and ePNP or ART as appropriate within 7 days of life | 7 days
  All infants enrolled in the study: 1) assessed for high-risk criteria for VHT at birth, 2) if high-risk, receiving enhanced post-natal prophylaxis (ePNP) and PoC birth EID testing, AND 3) if HIV-positive, initiated on ART

SECONDARY OUTCOMES:
Turnaround times for EID testing at birth, 4-6 weeks, and 14 weeks (time from sample collection to receipt of results by the health facility and communication of results to the mother/caregiver) and maternal PoC VL testing at delivery and 14 weeks | 14 weeks
Proportion and rate of VHT at birth, week 4-8, and week 14 | 14 weeks
Risk-factors associated with VHT | 14 weeks
  Demographic, socio-economic, and behavioral data collected from mothers
Adherence to PNP and ePNP | 14 weeks
Proportion and rate of clinical endpoints (mortality, morbidity) among HIV-positive infants at week 14, month 6, and month 12 | 12 months
Age at ART initiation among HIV-positive infants | 12 months
Risk factors for poor ART adherence among high-risk mothers and infants | 12 months
Proportion of HIV-positive infants virally suppressed at week 14, month 6, and month 12 | 12 months
Risk factors for poor viral suppression among HIV-positive infants | 12 months
Proportion of HIV-positive infants on ART that experience grade III or greater laboratory ART toxicity | 12 months
Retention to HIV EID and infant health care services | 14 weeks (Cohort A), 1 year (Cohort B)
Proportion of pregnant women presenting with criteria considered high-risk for VHT at delivery | 7 days
Proportion of mothers virally suppressed at week 14 post-partum | 14 weeks
Proportion and rate of post-partum mothers newly fulfilling high-risk criteria based on socio-behavioural criteria (i.e., adherence issues) | 14 weeks
Characteristics of transmitted viral strains (lineages, subtypes, resistance mutations) among HIV-positive infants and in comparison to their mothers viral sequences | 12 months
  Mother-child comparative genomic analysis and virus quasi-species diversity (major/minor and transmitted strains)
Proportion of HIV-positive infants who develop acquired drug resistance mutations during the study | 12 months
Characteristics of infant and maternal HIV strains to be neutralized against a panel of known broadly neutralizing antibody candidates (e.g., VRC07, 10-1074) and maternal autologous antibodies at time of transmission | 12 months
Average public healthcare and healthcare-related expenditures | 12 months
Average health worker time needed to care for mothers and infants per clinic visit, including for enhanced counselling sessions | 12 months
Cost per HIV-exposed infant fulfilling the primary outcome | 12 months
Empirical cost-effectiveness (incremental cost-effectiveness ratio) relating intervention costs to life-years saved among HIV-positive infants | 12 months
Average global and dimensional patient satisfaction | 14 weeks

OTHER OUTCOMES:
Hub-and-spoke model and provider satisfaction (health care personnel, focal point persons, counsellor) | 12 months
Socio-behavioural and personal aspects related to high-risk criteria for mother-child pairs (adherence, retention, disclosure, emotional well-being and health care satisfaction) | 14 weeks
Descriptions of tasks, functions, acceptability, challenge and workloads related to PVHT and neonatal HIV focal persons | 12 months
Descriptions of tasks, functions, acceptability, challenge and workloads related to counsellors (enhanced high-risk counselling) | 12 months
Description on eHealth functionality, satisfaction, acceptance of linkage procedures | 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- Centro de Investigacao Operacional de Beira (CIOB), Instituto Nacional de Saúde (INS), Ministério da Saúde,, Beira, Mozambique
- National Institute for Medical Research (NIMR), Mbeya, Mbeya, Tanzania

IPD SHARING:
Plan to Share IPD: No